CLINICAL TRIAL: NCT00497484
Title: Evaluation of rhGH Replacement Therapy in Patients With Pseudohypoparathyroidism Type Ia (PHP Ia)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Milan (Other)
Collaborators: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHP-IA-rhGH
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-06

CONDITIONS: Pseudohypoparathyroidism; Growth Hormone Deficiency, Dwarfism
MeSH Terms: conditions — Pseudohypoparathyroidism; Dwarfism, Pituitary

INTERVENTIONS:
Drug: recombinant human somatotropin

SUMMARY:
We have recently demonstrated resistance to GHRH leading to GH deficiency in patients with Pseudohypoparathyroidism type Ia (Mantovani et al., J Clin Endocrinol Metab, 2003. 88: 4070-4074). The purpose of this study is to evaluate the effect of at least 1-year GH replacement in these patients. In particular, we will focus our attention on growth velocity in children affected with this disease.

DETAILED DESCRIPTION:
Albright's Hereditary Osteodystrophy is a rare autosomal dominant disease characterized by a constellation of physical features including short stature, central obesity, round face, brachydactyly, subcutaneous calcifications and mental retardation. In the same family, it may present associated to end organ resistance to the action of different hormones, primarily PTH, TSH and gonadotropins and in this case it is named PHP type Ia, or on the contrary we may find it as an isolated defect and this is the case of PPHP.

In about 80% of affected families, heterozygous loss of function mutations in the Gs alpha gene are detected. It is of interest mutations inherited from the mother always lead to the complete form of the disorder, that is PHP; on the contrary when the same mutations are inherited from the father, patients show the physical abnormalities of Albright's Osteodystrophy, without any evidence of hormone resistance. This pattern of inheritance is consistent with a tissue-specific paternal imprinting of the Gs alpha gene. Imprinting is an epigenetic phenomenon by which one of the 2 alleles undergoes partial or total loss of expression; in the case of the Gs alpha gene one would expect that only the paternal allele should be lost in specific endocrine tissues, such as the kidney, the thyroid and the gonad, which are the target organs resistant to hormone action in PHP Ia. Indeed, our group demonstrated that in specific human endocrine tissues also Gs alpha transcription mainly derives from the maternal allele (Mantovani et al., J Clin Endocrinol Metab, 2002. 87: 4736-4740). In particular a predominant maternal origin of transcription was found in thyroid and gonad and these data are consistent with the clinical finding of TSH and gonadotropin resistance present in patients affected with PHP. Interestingly, we observed a predominance of the maternal allele also in the pituitary gland, an organ which is not classically included among the target organs resistant to hormone action in PHP Ia.

Following this observation, we have recently demonstrated resistance to GHRH leading to GH deficiency in most of our patients with PHP Ia (Mantovani et al., J Clin Endocrinol Metab, 2003. 88: 4070-4074). The purpose of this study is to evaluate the effect of at least 1-year GH replacement in these patients. In particular, we will focus our attention on growth velocity in children affected with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or genetic diagnosis of Pseudohypoparathyroidism type Ia
* Growth hormone deficiency

Exclusion Criteria:

* Known malignancies

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

PRIMARY OUTCOMES:
growth velocity | One year

SECONDARY OUTCOMES:
IGF-1 levels | one month

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Beck-Peccoz, MD/PhD, Study Director — Endocrine Unit, Dpt. of Medical Sciences, Fondazione Policlinico IRCCS, Milan
Locations (1):
- Endocrine Unit, Dpt. of Medical Sciences, Fondazione Policlinico IRCCS, Milan, Italy

REFERENCES:
- [Background] Mantovani G, Maghnie M, Weber G, De Menis E, Brunelli V, Cappa M, Loli P, Beck-Peccoz P, Spada A. Growth hormone-releasing hormone resistance in pseudohypoparathyroidism type ia: new evidence for imprinting of the Gs alpha gene. J Clin Endocrinol Metab. 2003 Sep;88(9):4070-4. doi: 10.1210/jc.2002-022028. PMID 12970263
- [Background] Germain-Lee EL, Groman J, Crane JL, Jan de Beur SM, Levine MA. Growth hormone deficiency in pseudohypoparathyroidism type 1a: another manifestation of multihormone resistance. J Clin Endocrinol Metab. 2003 Sep;88(9):4059-69. doi: 10.1210/jc.2003-030028. PMID 12970262
- [Derived] Mantovani G, Ferrante E, Giavoli C, Linglart A, Cappa M, Cisternino M, Maghnie M, Ghizzoni L, de Sanctis L, Lania AG, Beck-Peccoz P, Spada A. Recombinant human GH replacement therapy in children with pseudohypoparathyroidism type Ia: first study on the effect on growth. J Clin Endocrinol Metab. 2010 Nov;95(11):5011-7. doi: 10.1210/jc.2010-1649. Epub 2010 Aug 18. PMID 20719837